CLINICAL TRIAL: NCT06587555
Title: Correlations Between Symptoms of Anxiety And/or Depression with Dysphagia Severity Level
Status: Not yet recruiting | Type: Observational
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Principal Investigator, Vitriana Biben, Dr. Vitriana Biben, dr., Sp.K.F.R, NM(K), Universitas Padjadjaran
Other Study IDs: IKFR-202408.02
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Dysphagia; Anxiety; Depression
Keywords: Dysphagia Severity Level; Anxiety; Depression; Dyspahgia; HADS
MeSH Terms: conditions — Deglutition Disorders; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to know any CORRELATIONS BETWEEN SYMPTOMS OF ANXIETY AND / OR DEPRESSION WITH DYSPHAGIA SEVERITY LEVEL in is all of the new or ongoing patients with dysphagia in the Neurorehabilitation Department at Hasan Sadikin General Hospital Bandung and who meet the inclusion and exclusion criteria. The main questions it aims to answer are:

Hypothesis 1 H0 : There is no correlation between increased severity of dysphagia and higher levels of anxiety symptoms H1 : There is a correlation between increased severity of dysphagia and higher levels of anxiety

Hypothesis 2 H0 : There is no correlation between increased severity level of dysphagia and higher level of depression symptoms H1 : There is a correlation between increased severity of dysphagia and higher levels of depression

Hypothesis 3 H0 : There is no correlation between increased severity level of anxiety and dysphagia and higher level of depression symptoms H1 : There is a correlation between increased severity of anxiety and dysphagia and higher levels of depression

DETAILED DESCRIPTION:
This study is an analytical observational study with a cross-sectional design, then correlation analysis was carried out, to analyse the correlation between Severity level of dysphagia with anxiety and / or depression. This Study performed at Hasan Sadikin Hospital between August 2024 - March 2025

Study Subject : The target population for this study is all of the new or ongoing patients with dysphagia in the Neurorehabilitation Department at Hasan Sadikin General Hospital Bandung and who meet the inclusion and exclusion criteria.

Inclusion criteria :

* Participants aged 18 years and above.
* Individuals diagnosed with dysphagia by a qualified healthcare professional
* Participants with documented anxiety and/or depression symptoms were assessed using standardized psychological assessments
* Willing to participate

Exclusion criteria :

Participants who have MOCA INA < 18 Participants with severe malnutrition, showed by BMI WHO Asia Pacific < 18.5 Participants with unstable hemodynamics, GCS < 15 Participants who had a history of diagnosed anxiety and / or depression Participants who had a history of using an antipsychotic drug

Sample Size Determination :

The sample size in this study was determined using correlation analysis, to see the correlation between variables, with a minimum number of samples of 30 research subjects obtained.

Confounding Factors :

1. Underlying disease
2. Age
3. Duration of Rehabilitation Therapy
4. Type of Rehabilitation Theraphy

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18 years and above.
2. Individuals diagnosed with dysphagia by a qualified healthcare professional
3. Participants with documented anxiety and/or depression symptoms were assessed using standardized psychological assessments
4. Willing to participate

Exclusion Criteria:

1. Participants who have MOCA INA < 18
2. Participants with severe malnutrition, showed by BMI WHO Asia Pacific < 18.5
3. Participants with unstable hemodynamics, GCS < 15
4. Participants who had a history of diagnosed anxiety and / or depression
5. Participants who had a history of using an antipsychotic drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for this study is all of the new or ongoing patients with dysphagia in the Neurorehabilitation Department at Hasan Sadikin General Hospital Bandung and who meet the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety and / or Depression Symptoms Measure using HADS questionary | September 2024 - January 2025
  Hospital Anxiety and Depression Questionnaire (HADS) are ranging from 0-7 points meaning no depression/ anxiety cases (ie, non- cases), 8-10 points representing borderline or doubtful cases, and ≥11 points suggesting anxiety or depressive cases

CONTACTS AND LOCATIONS:
Overall Officials: Vitriana Biben, Study Director — University Padjajaran
Locations (1):
- Hasan Sadikin General Hospital, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Matsuo K, Palmer JB. Anatomy and physiology of feeding and swallowing: normal and abnormal. Phys Med Rehabil Clin N Am. 2008 Nov;19(4):691-707, vii. doi: 10.1016/j.pmr.2008.06.001. PMID 18940636
- [Background] Kwon S, Cha S, Kim J, Han K, Paik NJ, Kim WS. Trends in the incidence and prevalence of dysphagia requiring medical attention among adults in South Korea, 2006-2016: A nationwide population study. PLoS One. 2023 Jun 28;18(6):e0287512. doi: 10.1371/journal.pone.0287512. eCollection 2023. PMID 37379287
- [Background] Kim DY, Park HS, Park SW, Kim JH. The impact of dysphagia on quality of life in stroke patients. Medicine (Baltimore). 2020 Aug 21;99(34):e21795. doi: 10.1097/MD.0000000000021795. PMID 32846813
- [Background] Bendsen BB, Jensen D, Westmark S, Krarup AL, Riis J, Melgaard D. The Quality of Life in Citizens with Oropharyngeal Dysphagia-A Cross-Sectional Study. J Clin Med. 2022 Jul 20;11(14):4212. doi: 10.3390/jcm11144212. PMID 35887975
- [Background] Bushuven S, Niebel I, Huber J, Diesener P. Emotional and Psychological Effects of Dysphagia: Validation of the Jugendwerk Dysphagia Emotion and Family Assessment (JDEFA). Dysphagia. 2022 Apr;37(2):375-391. doi: 10.1007/s00455-021-10289-1. Epub 2021 Apr 4. PMID 33817751
- [Background] Brenes GA. Anxiety, depression, and quality of life in primary care patients. Prim Care Companion J Clin Psychiatry. 2007;9(6):437-43. doi: 10.4088/pcc.v09n0606. PMID 18185823
- [Background] Verdonschot RJ, Baijens LW, Serroyen JL, Leue C, Kremer B. Symptoms of anxiety and depression assessed with the Hospital Anxiety and Depression Scale in patients with oropharyngeal dysphagia. J Psychosom Res. 2013 Nov;75(5):451-5. doi: 10.1016/j.jpsychores.2013.08.021. Epub 2013 Sep 3. PMID 24182634
- [Background] Krekeler BN, Broadfoot CK, Johnson S, Connor NP, Rogus-Pulia N. Patient Adherence to Dysphagia Recommendations: A Systematic Review. Dysphagia. 2018 Apr;33(2):173-184. doi: 10.1007/s00455-017-9852-9. Epub 2017 Sep 30. PMID 28965240
- [Background] Doruk C, Mocchetti V, Rives H, Christos P, Rameau A. Correlations Between Anxiety and/or Depression Diagnoses and Dysphagia Severity. Laryngoscope. 2024 May;134(5):2115-2120. doi: 10.1002/lary.31164. Epub 2023 Nov 9. PMID 37942834
- [Background] DiMatteo MR, Lepper HS, Croghan TW. Depression is a risk factor for noncompliance with medical treatment: meta-analysis of the effects of anxiety and depression on patient adherence. Arch Intern Med. 2000 Jul 24;160(14):2101-7. doi: 10.1001/archinte.160.14.2101. PMID 10904452
- [Background] Adkins C, Takakura W, Spiegel BMR, Lu M, Vera-Llonch M, Williams J, Almario CV. Prevalence and Characteristics of Dysphagia Based on a Population-Based Survey. Clin Gastroenterol Hepatol. 2020 Aug;18(9):1970-1979.e2. doi: 10.1016/j.cgh.2019.10.029. Epub 2019 Oct 24. PMID 31669055
- [Background] Karisik A, Dejakum B, Moelgg K, Komarek S, Toell T, Mayer-Suess L, Pechlaner R, Kostner S, Sollereder S, Kiechl S, Rossi S, Schoenherr G, Lang W, Kiechl S, Knoflach M, Boehme C; STROKE-CARD Registry study group. Association between dysphagia and symptoms of depression and anxiety after ischemic stroke. Eur J Neurol. 2024 May;31(5):e16224. doi: 10.1111/ene.16224. Epub 2024 Feb 2. PMID 38308469
- [Background] Tanaka M, Szabo A, Vecsei L. Integrating Armchair, Bench, and Bedside Research for Behavioral Neurology and Neuropsychiatry: Editorial. Biomedicines. 2022 Nov 22;10(12):2999. doi: 10.3390/biomedicines10122999. PMID 36551755
- [Background] Mori T, Wakabayashi H, Kishima M, Itoda M, Fujishima I, Kunieda K, Ohno T, Shigematsu T, Oshima F, Ogawa N, Nishioka S, Momosaki R, Shimizu A, Saito Y, Yamada M, Ogawa S. Association between Inflammation and Functional Outcome in Patients with Sarcopenic Dysphagia. J Nutr Health Aging. 2022;26(4):400-406. doi: 10.1007/s12603-022-1769-9. PMID 35450997
- [Background] Li Y, Hu N, Yang D, Oxenkrug G, Yang Q. Regulating the balance between the kynurenine and serotonin pathways of tryptophan metabolism. FEBS J. 2017 Mar;284(6):948-966. doi: 10.1111/febs.14026. Epub 2017 Feb 20. PMID 28118532
- [Background] Nguyen NP, Vos P, Karlsson U, Nguyen P, Dutta S, Lemanski C, Ludin A, Rose S, Nguyen LM, Ward H, Huang S, Sallah S. Quality of life following chemoradiation and postoperative radiation for locally advanced head and neck cancer. ORL J Otorhinolaryngol Relat Spec. 2007;69(5):271-6. doi: 10.1159/000103870. Epub 2007 Jun 12. PMID 17565229
- [Background] Tiksnadi BB, Triani N, Fihaya FY, Turu' Allo IJ, Iskandar S, Putri DAE. Validation of Hospital Anxiety and Depression Scale in an Indonesian population: a scale adaptation study. Fam Med Community Health. 2023 Jun;11(2):e001775. doi: 10.1136/fmch-2022-001775. PMID 37277187
- [Background] Soares-Filho GL, Freire RC, Biancha K, Pacheco T, Volschan A, Valenca AM, Nardi AE. Use of the hospital anxiety and depression scale (HADS) in a cardiac emergency room: chest pain unit. Clinics (Sao Paulo). 2009;64(3):209-14. doi: 10.1590/s1807-59322009000300011. PMID 19330247
- [Background] Dziewas R, Auf dem Brinke M, Birkmann U, Brauer G, Busch K, Cerra F, Damm-Lunau R, Dunkel J, Fellgiebel A, Garms E, Glahn J, Hagen S, Held S, Helfer C, Hiller M, Horn-Schenk C, Kley C, Lange N, Lapa S, Ledl C, Lindner-Pfleghar B, Mertl-Rotzer M, Muller M, Neugebauer H, Ozsucu D, Ohms M, Perniss M, Pfeilschifter W, Plass T, Roth C, Roukens R, Schmidt-Wilcke T, Schumann B, Schwarze J, Schweikert K, Stege H, Theuerkauf D, Thomas RS, Vahle U, Voigt N, Weber H, Werner CJ, Wirth R, Wittich I, Woldag H, Warnecke T. Safety and clinical impact of FEES - results of the FEES-registry. Neurol Res Pract. 2019 Apr 26;1:16. doi: 10.1186/s42466-019-0021-5. eCollection 2019. PMID 33324882
- [Background] Farooq N, Khatoon S, Malik AN, Rathore FA. Role of Vitalstim(R) In The Management Of Patients With Dysphagia: A MiniReview. J Pak Med Assoc. 2023 Jun;73(6):1346-1348. doi: 10.47391/JPMA.23-46. PMID 37427651
- [Background] Liang Y, Lin J, Wang H, Li S, Chen F, Chen L, Li L. Evaluating the Efficacy of VitalStim Electrical Stimulation Combined with Swallowing Function Training for Treating Dysphagia following an Acute Stroke. Clinics (Sao Paulo). 2021 Nov 8;76:e3069. doi: 10.6061/clinics/2021/e3069. eCollection 2021. PMID 34755758
- [Background] Tan Z, Wei X, Tan C, Wang H, Tian S. Effect of neuromuscular electrical stimulation combined with swallowing rehabilitation training on the treatment efficacy and life quality of stroke patients with dysphagia. Am J Transl Res. 2022 Feb 15;14(2):1258-1267. eCollection 2022. PMID 35273727
- See also: World Health Organization. Anxiety disorders — https://www.who.int/news-room/fact-sheets/detail/anxiety-disorders